CLINICAL TRIAL: NCT02782260
Title: Assessment of the Efficacy of Ocular Dipyridamole in the Treatment of Dry Eye Symptomology in Subjects With Pterygium
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ariel University (Other)
Responsible Party: Principal Investigator, Lily Karmona, Dr, Ariel University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0064-16-WOMC
Record Dates: First submitted 2016-05-10; First posted 2016-05-25 (Estimated); Last update posted 2016-05-25 (Estimated); Status verified 2016-05

CONDITIONS: Dry Eye Syndromes; Pterygium
MeSH Terms: conditions — Dry Eye Syndromes; Pterygium | interventions — Dipyridamole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Experimental): Dipyridamole eye drops 8.48 mg in 100ml
  1 drop three times a day for 1 year
  Interventions: Drug: Dipyridamole
- Placebo (Placebo Comparator): Fluorescein in Active Vehicle
  1 drop three times a day for 1 year
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dipyridamole
  Arms: Active
Drug: Placebo
  Arms: Placebo

SUMMARY:
Subjects with pterygium and associated dry eye symptoms (DES) are randomized into an active cohort (receiving ocular administration of Dipyridamole) or placebo cohort (ocular administration of vehicle). Monthly follow up is conducted for 12 months. Testing conducted at follow up will assess dry eye / pterygium symptoms and endpoints and review the efficacy of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent.
* Ineligible or refused surgical excision, or had recurrence of pterygium following surgical excision
* Able to follow the study instructions, including application of the study product
* Agreement not to change the type of lubricating eye drops used (if any) during their participation in the study.
* Assessed as having at least pterygium stage 0-1 (pinguecula) based on Johnston, Williams & Sheppard's classification for pterygium
* Concomitant dry eye symptoms, as determined by one or more of the following Subject interview (modified Ocular Surface Disease Index test), Tearing, Itch / foreign body sensation, Positive Fluorescein test, Positive TBUT test, Positive Tear meniscus test

Exclusion Criteria:

* Inability to provide informed consent
* Dry eye due to other factors
* Known lacrimal obstruction
* Contact lens wearers
* Non-corrected refraction
* Allergy or sensitivity to dipyridamole or excipients
* Use of dipyridamole in the last 6 months
* Other eye conditions (i.e. active ocular infection, herpes keratitis in last 6 months, corneal disorder abnormality excluding pterygium, history of ocular acne rosacea, blepharitis) which would impact results
* Diagnosis of ALS (Amyotrophic lateral sclerosis)
* Existing conditions which are contraindicated or precaution in use of dipyridamole or excipients
* Use of eye drops (other than ocular lubricants)
* Pregnant or breastfeeding
* Inability to apply the medical product or follow the study procedures
* Anything that the PI thinks would impact the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-10 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Assess the changes in dry eye parameters via a change in tear secretion rate | 6 months
  Change in the tear secretion rate will be defined by successful change in parameters of ONE of the following testing methods compared to baseline:
  1. Fluorescein - Improvement of one of the quadrants sufficient to change the severity rating
  2. TBUT (Tear Breakup time) - Decreased by at least 1 second
  3. Tear meniscus test - Increase of at least 0.2mm
Assess the changes in dry eye parameters via reduction in dry eye symptomology. | 6 months
  Reduction in dry eye symptomology will be defined as ONE of the following relative to baseline, determined by subject feedback
  * An improvement in questionnaire scores
  * Specified improvement in blurred vision grading
  * Specified improvement in tearing grading
  * Specified improvement in itch / foreign body (grittiness) sensation grading.

SECONDARY OUTCOMES:
A minimum significant reversion of pterygia relative to baseline or cessation of growth of pterygium | 12 months
  Minimum significant reversion will be defined as a decrease in vascularisation, or a measurable decrease from baseline of OCT (Ocular Coherence Tomography) measured parameters (height or width).

IPD SHARING:
Plan to Share IPD: Undecided